CLINICAL TRIAL: NCT02211573
Title: Effects of Aquatic Aerobic Training on Body Composition and Cardiorespiratory and Metabolic Variables in Patients With Coronary Artery Disease
Brief Title: Aquatic Aerobic Training, Cardiorespiratory and Metabolic Variables in Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Responsible Party: Principal Investigator, Elie Fiogbé, Professor, Universidade Metodista de Piracicaba
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03/14
Record Dates: First submitted 2014-08-05; First posted 2014-08-07 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Arteriosclerosis, Coronary
Keywords: Autonomic Nervous System, Body composition, Oxygen Uptake,; Water Based Physical Training.
MeSH Terms: conditions — Coronary Artery Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Patients of this group don't performed physical training
- Exercise, Aerobic (Water based) (Experimental): Patients of this group were submitted to an aerobic water based physical training
  Interventions: Other: Exercise, Aerobic (Water based)

INTERVENTIONS:
Other: Exercise, Aerobic (Water based) — Patients of this group were submitted to an aerobic water based physical training
  Arms: Exercise, Aerobic (Water based)

SUMMARY:
Although approaches to reduce cardiovascular disease, coronary artery disease (CAD) remains the leading cause of mortality in the industrialized world. In order to reduce the deleterious effects of the atherosclerotic process, proposals for non-pharmacological treatment have been used, such as cardiac rehabilitation programs, with emphasis on exercise -based therapy. Traditionally aerobic exercises like biking, walking and jogging are conducted, however, alternative ways such as aquatic exercise training have been proposed, however, the cardiorespiratory adaptations in this population are not well documented in the literature. Thus, the aim of this study was to evaluate the effects of aquatic aerobic training (AAT) on body composition, autonomic modulation of heart rate (HR) and cardiorespiratory and metabolic variables in patients with CAD. This was a longitudinal clinical trial with a sample allocated for convenience, in which twenty-one patients were male, with a diagnosis of CAD, which were divided into control group (CG were studied, n=8), who was only assessed, and training group (TG, n=13). All patients underwent assessment of body composition, heart rate variability (HRV) at rest in the supine posture, and cardiopulmonary exercise testing (CPET), performed before and after the AAT program. The training protocol consisted of three sessions per week on alternate days for 16 weeks, totaling 48 sessions, which had lasted approximately one hour. The exercise intensity was prescribed between 80 and 110% of the first ventilatory threshold (VT1) obtained in CPET. Given that these parameters represent risk markers for cardiovascular events in the population studied, the results suggest that the AAT proposed in this study may be an important therapeutic strategy to be incorporated into cardiac rehabilitation programs.

DETAILED DESCRIPTION:
1. Personal Data recording:

   * History: personal data, lifestyle and food, family history, current and previous history of disease.
   * Physical examination: cardiac and lung auscultation,measurement of heart rate (HR), blood pressure (BP), body weight and height.
2. Assessments:

   All experimental procedures were performed in the morning in order to minimize the influence of circadian cycle. The temperature of the experimental room was maintained between 22 ° C and 24 ° C with relative humidity between 40% and 60%. Patients were familiarized with the experimental protocol, and instructed not to ingest stimulant drinks such as coffee, tea and soft drinks, do not drink alcohol, do not perform strenuous exercise (48 hours before surgery), and to perform a light meal at least four hours before the collections.

   Aiming to verify if the baseline conditions were suitable for the beginning of the experimental procedures, the patients remained 15 minutes of rest in the supine position, and recorded blood pressure (BP) and HR.

   After this, were performed:
   * Analysis of body composition by bioelectrical impedance analysis.
   * Registration of HR and NN intervals (NN) during rest, in the supine and sitting positions.
   * Recording of HR and NN during rest in the supine position, sitting, standing and during respiratory sinus arrhythmia maneuver.
   * Spirometric test and
   * Cardiopulmonary exercise test (CPET). This is a submaximal CPET performed on a treadmill, in order to verify and identify possible changes in hemodynamic, electrocardiographic induced to physical exertion, their aerobic functional capacity as well as to prescribe physical training protocol.
3. Training:

   After this assessment the volunteers were trained by a aerobic water based physical training program for 4 weeks.
4. Second assessment:

Components of the first assessment have been repeated at the end of each month of physical training.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis by angiography
* sedentaries
* family story of cardiac disease
* obesity

Exclusion Criteria:

* frequent arrhythmias at rest
* triggered by physical effort
* unstable angina
* chronic obstructive pulmonary disease
* insulin-dependent diabet
* renal failure
* sequel of stroke
* uncontrolled hypothyroidism
* water phobia
* skin infections, allergic reactions to chlorine,
* urinary incontinence and
* musculoskeletal and neuromuscular disorders precluding physical tests and training sessions

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-05; Primary Completion 2013-10 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in autonomic system modulation | baseline and 16 weeks
  Change in autonomic system modulation in assess by comparing the heart rate variability at baseline and after a 16 weeks of aerobic water and land based physical training.

SECONDARY OUTCOMES:
Change in body composition | baseline and 16 weeks
  Change in body composition is assess by comparing the body composition at baseline and after a 16 weeks of aerobic water and land based physical training.

OTHER OUTCOMES:
Oxygen uptake | 16 Weeks
  Change in oxygen uptake is assessed by comparing the oxygen uptake at baseline and after a 16 weeks of aerobic water and land based physical training.

CONTACTS AND LOCATIONS:
Overall Officials: Elie Fiogbé, Ms, Principal Investigator — Universidade Metodista de Piracicaba
Locations (1):
- Universidade Metodista de Piracicaba, Piracicaba, São Paulo, Brazil